CLINICAL TRIAL: NCT00546949
Title: Treatment of Lumbar Spinal Stenosis; Comparison of Two Different Surgical Methods; Mini-Invasive Decompression to X-Stop (LSSS)
Brief Title: Treatment of Lumbar Spinal Stenosis; Comparison of Two Different Surgical Methods; Mini-invasive Decompression to X-stop
Acronym: LSSS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: analysis at 50% inclusion showed 4 times larger reoperation rate in X-stop group
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSSL-16279
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Lumbar Spinal Stenosis; Radiculopathy
Keywords: Decompression, Surgical; x-stop; lumbar decompression; spinal stenosis; radiculopathy
MeSH Terms: conditions — Spinal Stenosis; Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- decompression (Active Comparator): Minimal invasive decompression
  Interventions: Procedure: Minimal invasive decompression
- x-stop (Experimental): X-stop, an interspinous decompression device
  Interventions: Procedure: Interspinous Process Decompression (IPD)

INTERVENTIONS:
Procedure: Minimal invasive decompression — foraminotomy, laminotomy, microscopic decompression
  Other Names: mini-invasive decompression
  Arms: decompression
Procedure: Interspinous Process Decompression (IPD) — Interspinous device
  Other Names: X-stop
  Arms: x-stop

SUMMARY:
The purpose of this study is to compare two surgery methods on lumbar spinal stenosis: minimal invasive decompression and X-stop. It is a prospective randomized multicenter study including patients with lumbar spinal stenosis on one or two levels, and neurogenic intermittent claudication. Effect assessment will include measures of pain and self-evaluated health condition, a full economical evaluation, and areal measurements (MR imaging and roentgen analyses)

ELIGIBILITY:
Inclusion Criteria:

* neurogenic intermittent claudication due to lumbar spinal stenosis
* diagnosed on MRI in maximum two levels
* walking distance on 250 metres
* symptom relief on flexion of the lumbar spine
* duration of the symptoms more than 6 months
* non-operative treatment is tried or considered as not indicated

Exclusion Criteria:

* vascular claudicatio intermittens
* spinal stenosis on more than 2 levels
* cauda equina syndrome
* severe paresis
* clinical monoradiculopathy
* grave scoliosis
* previous lumbar surgery
* degenerative spondylolisthesis more than 25%
* spondylolysis with listhesis
* osteoporotic fracture in lumbal column
* clinical and radiological (both) arthritis in the hip joint
* ASA >3
* verified polyneuropathy on neurophysiological test

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2007-03; Primary Completion 2011-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Claudication | 2 years
  Zürich Claudication Questionnaire

SECONDARY OUTCOMES:
self-evaluated health condition | 2 years
  SF36, Oswestry Disability Index (ODI), EQ5-D and VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Greger Lønne, MD, Principal Investigator — Norwegian University of Sciense and Technology
Locations (1):
- Nastional Senter for Spinal Disorders, Trondheim, Norway

REFERENCES:
- [Result] Lonne G, Johnsen LG, Rossvoll I, Andresen H, Storheim K, Zwart JA, Nygaard OP. Minimally invasive decompression versus x-stop in lumbar spinal stenosis: a randomized controlled multicenter study. Spine (Phila Pa 1976). 2015 Jan 15;40(2):77-85. doi: 10.1097/BRS.0000000000000691. PMID 25575084
- [Result] Lonne G, Johnsen LG, Aas E, Lydersen S, Andresen H, Ronning R, Nygaard OP. Comparing cost-effectiveness of X-Stop with minimally invasive decompression in lumbar spinal stenosis: a randomized controlled trial. Spine (Phila Pa 1976). 2015 Apr 15;40(8):514-20. doi: 10.1097/BRS.0000000000000798. PMID 25608246